CLINICAL TRIAL: NCT01658683
Title: Ecologically Optimizing Exercise Maintenance in Men and Women Post-Cardiac Rehabilitation: A Randomized Controlled Trial of Efficacy With Economics
Brief Title: The Efficacy and Economics of Exercise Maintenance Post-Cardiac Rehabilitation
Acronym: ECOPCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201200579-01
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Cardiac Rehabilitation; Exercise Maintenance; Facilitator; Managed Home Exercise; Community Based Exercise
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Facilitator Intervention (Experimental): The intervention employs small group counseling teleconferences (5),personal telephone contacts (3) and community Heart Wise Exercise program demonstrations.
  Interventions: Behavioral: Exercise Facilitator Intervention
- Usual Care (No Intervention): Usual care for cardiac rehab graduates provided by the University of Ottawa Heart Institute Minto Prevention & Rehabilitation Centre and the Cardiovascular Rehabilitation and Prevention Centre at the University Health Network.

INTERVENTIONS:
Behavioral: Exercise Facilitator Intervention — The 50 week intervention includes 5 small group counseling teleconferences, 3 personal telephone calls and Heart Wise Exercise program demonstrations. During the teleconferences and personal telephone calls, the facilitator discusses the importance of exercise. Participants review their activity diaries, identify barriers to exercise maintenance experienced to date and brainstorm solutions as a group. In addition, the facilitator conducts community program demonstrations at Heart Wise Exercise program locations in Ottawa and Toronto for interested participants.
  Arms: Exercise Facilitator Intervention

SUMMARY:
The purpose of this study is to develop a new intervention to improve the transition of patients from structured, supervised exercise to self-managed home- or approved community-based exercise programs in an effort to increase maintenance of exercise behaviour post cardiac rehabilitation (CR). The goal of the study is that those receiving the intervention will engage in at least 30 minutes of physical activity at a moderate or vigorous intensity 5 or more days per week, 26, 52 and 78 weeks after CR compared to those in the usual care group. The new intervention will be delivered by trained exercise facilitators (physiotherapists or exercise specialists) and will make use of: small group counseling teleconferences (5 sessions); personal telephone contacts (3 sessions), and community program demonstrations that would facilitate linkages between patients and approved community programs known as Heart Wise Exercise programs available in Ottawa and Toronto. The trial will be conducted at the Minto Prevention and Rehabilitation Centre at the University of Ottawa Heart Institute and the Cardiovascular Rehabilitation and Prevention Centre at the University Health Network (Peter Munk Cardiac Centre [PMCC] and Toronto Rehabilitation Institute [TRI]) sites. The study has a target enrollment of 604 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently participating in an on-site CR program of ≥ 8-week duration (to ensure that outcomes are not confounded by exposure to home-based or telephone-based case managed programs)
* Patient has graduated from CR (to ensure that the study is evaluating an intervention to help sustain and improve maintenance of exercise behaviour
* Patient has a documented diagnosis of CAD (to ensure homogeneity of the patient population)
* Patient is 18 years of age or older
* Patient is able and willing to provide informed consent
* Able to walk unaided at 2 mph

Exclusion Criteria:

* Patient has New York Heart Association class III or IV heart failure (because this might interfere with the ability to achieve recommended exercise levels and to ensure homogeneity of the patient population)
* Patient is pregnant, lactating or planning to become pregnant during the study period (because this might interfere with the ability to achieve recommended exercise levels)
* Patient is unable to read and understand English or French
* Planning to leave the province or region in the next 12 months
* Member of the participant's household is already participating in the study
* The participant is unable, in the opinion of the qualified investigator, to participate in unsupervised exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
9-day accelerometer-measured physical activity of moderate and vigorous intensity | 78 weeks
  Physical activity will be measured directly by having participants wear the Actigraph GT3X accelerometer (Actigraph, Pensacola, Florida) over the right hip for a 9-day recording period, excluding periods when they are sleeping, swimming, or bathing. The activity monitor provides measurements including activity counts, energy expenditure, and step counts, in addition to activity intensity levels. Participants will be considered to be maintaining exercise at guideline recommended levels if they undertake ≥ 30 minutes of moderate and/or vigorous intensity physical activity on ≥ five days.

SECONDARY OUTCOMES:
Symptom limited graded exercise test with electrocardiographic monitoring using a ramp protocol on a treadmill | 52 weeks
  A random sub-sample of participants (N = 124) will complete a symptom limited graded exercise test with electrocardiographic monitoring using a ramp protocol on a treadmill at baseline and at 52 weeks. Exercise tolerance will also be assessed using the Duke Activity Status Index (DASI), a self-administered questionnaire that measures a patient's functional capacity and is used as an estimate of an individual's peak oxygen uptake
Quality of life measured by the the EuroQoL 5D | 78 weeks
  The EQ-5D is the current gold standard measure of generic quality of life, has been used in numerous studies and has been validated in many languages. The EQ-5D consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale. The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Cardiovascular risk factors measured by body mass index and blood pressure. | 78 weeks
  Height and weight is measured for the determination of body mass index (BMI). Waist circumference is measured using a non-stretchable standard tape measure. Systolic blood pressure is measured in a seated position after a five-minute rest period using an automated, non-invasive blood pressure monitor (BPTru) that automatically performs six measurements
Enrollment in Heart Wise Exercise programs | 78 weeks
  Enrollment in community-based and Heart Wise Exercise programs will be queried in the follow-up surveys.
Mediators of Intervention Effect | 78 weeks
  1.Physical activity history 2.Physical activity self-regulation 3. Action planning 4. Intentions to exercise 5. Beliefs about the benefits of and barriers to exercise 5. Task self-efficacy 6. Barrier self-efficacy 7. Social support from family and friends 8. Autonomy support derived from health care providers 9. Home exercise equipment 10. Neighbourhood environmental attributes of walkability and access to recreation facilities 11. Adherence to medications
Cost-effectiveness and cost-utility | 78 weeks
  Health effects are measured by overall survival time; event-free time from myocardial infarction, revascularization or death; and quality adjusted life years. Participants are linked to health administrative data to allow health care utilization to be tracked. Participants complete a monthly diary to record time for counseling and physical activities, out-of-pocket expenses, and items related to productivity, including lost work days, home care expenses due to reduced function or cardiac disability. Data is collected on the resources expended for each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Reid, MBA, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation; Sherry Grace, PhD, Principal Investigator — Peter Munk Cardiac Centre; Andrew Pipe, MD, Study Chair — Ottawa Heart Institute Research Corporation; Caroline Chessex, MD, MSc, Study Chair — Peter Munk Cardiac Centre; Chris Blanchard, PhD, Study Chair — Dalhousie University; Murray Krahn, MD, MSc, Study Chair — University of Toronto, Toronto Health Economics and Technology Assessment Collaborative; Doug Manuel, MD, Study Chair — Institute for Clinical Evaluative Sciences; Kori Kingsbury, MSN, MPA, Study Chair — Cardiac Care Network of Ontario; Jennifer Harris, BSc, PT, Study Chair — Ottawa Heart Institute Research Corporation; Kerri-Anne Mullen, MSc, Study Chair — Institute for Clinical Evaluative Sciences; Amy Mark, PhD, Study Chair — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - York University and University Health Network, Toronto, Ontario

REFERENCES:
- [Background] Grace SL, Chessex C, Arthur H, Chan S, Cyr C, Dafoe W, Juneau M, Oh P, Suskin N. Systematizing Inpatient Referral to Cardiac Rehabilitation 2010: Canadian association of cardiac rehabilitation and Canadian cardiovascular society joint position paper. J Cardiopulm Rehabil Prev. 2011 May-Jun;31(3):E1-8. doi: 10.1097/HCR.0b013e318219721f. PMID 21460733
- [Background] Blanchard CM, Reid RD, Morrin LI, McDonnell L, McGannon K, Rhodes RE, Spence JC, Edwards N. Demographic and clinical determinants of moderate to vigorous physical activity during home-based cardiac rehabilitation: the home-based determinants of exercise (HOME) study. J Cardiopulm Rehabil Prev. 2010 Jul-Aug;30(4):240-5. doi: 10.1097/HCR.0b013e3181d0c4ae. PMID 20216322
- [Background] Reid RD, Morrin LI, Pipe AL, Dafoe WA, Higginson LA, Wielgosz AT, LeHaye SA, McDonald PW, Plotnikoff RC, Courneya KS, Oldridge NB, Beaton LJ, Papadakis S, Slovinec D'Angelo ME, Tulloch HE, Blanchard CM. Determinants of physical activity after hospitalization for coronary artery disease: the Tracking Exercise After Cardiac Hospitalization (TEACH) Study. Eur J Cardiovasc Prev Rehabil. 2006 Aug;13(4):529-37. doi: 10.1097/01.hjr.0000201513.13343.97. PMID 16874141
- [Background] Blanchard CM, Courneya KS, Rodgers WM, Fraser SN, Murray TC, Daub B, Black B. Is the theory of planned behavior a useful framework for understanding exercise adherence during phase II cardiac rehabilitation? J Cardiopulm Rehabil. 2003 Jan-Feb;23(1):29-39. doi: 10.1097/00008483-200301000-00007. PMID 12576910
- [Background] Reid RD, Dafoe WA, Morrin L, Mayhew A, Papadakis S, Beaton L, Oldridge NB, Coyle D, Wells GA. Impact of program duration and contact frequency on efficacy and cost of cardiac rehabilitation: results of a randomized trial. Am Heart J. 2005 May;149(5):862-8. doi: 10.1016/j.ahj.2004.09.029. PMID 15894969
- [Background] Bock BC, Carmona-Barros RE, Esler JL, Tilkemeier PL. Program participation and physical activity maintenance after cardiac rehabilitation. Behav Modif. 2003 Jan;27(1):37-53. doi: 10.1177/0145445502238692. PMID 12587259
- [Background] Izawa KP, Yamada S, Oka K, Watanabe S, Omiya K, Iijima S, Hirano Y, Kobayashi T, Kasahara Y, Samejima H, Osada N. Long-term exercise maintenance, physical activity, and health-related quality of life after cardiac rehabilitation. Am J Phys Med Rehabil. 2004 Dec;83(12):884-92. doi: 10.1097/01.phm.0000143404.59050.11. PMID 15624566
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Sallis JF, Kerr J, Carlson JA, Norman GJ, Saelens BE, Durant N, Ainsworth BE. Evaluating a brief self-report measure of neighborhood environments for physical activity research and surveillance: Physical Activity Neighborhood Environment Scale (PANES). J Phys Act Health. 2010 Jul;7(4):533-40. doi: 10.1123/jpah.7.4.533. PMID 20683096
- [Background] Shaw JW, Johnson JA, Coons SJ. US valuation of the EQ-5D health states: development and testing of the D1 valuation model. Med Care. 2005 Mar;43(3):203-20. doi: 10.1097/00005650-200503000-00003. PMID 15725977
- [Background] Heran BS, Chen JM, Ebrahim S, Moxham T, Oldridge N, Rees K, Thompson DR, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001800. doi: 10.1002/14651858.CD001800.pub2. PMID 21735386
- [Background] Hodges JM. Reflections: Occupational therapy. Am J Occup Ther. 1976 Aug;30(7):409-10. No abstract available. PMID 782256
- [Background] Izawa KP, Watanabe S, Omiya K, Hirano Y, Oka K, Osada N, Iijima S. Effect of the self-monitoring approach on exercise maintenance during cardiac rehabilitation: a randomized, controlled trial. Am J Phys Med Rehabil. 2005 May;84(5):313-21. doi: 10.1097/01.phm.0000156901.95289.09. PMID 15829777
- [Background] Johnson NA, Lim LL, Bowe SJ. Multicenter randomized controlled trial of a home walking intervention after outpatient cardiac rehabilitation on health-related quality of life in women. Eur J Cardiovasc Prev Rehabil. 2009 Oct;16(5):633-7. doi: 10.1097/HJR.0b013e32832e8eba. PMID 19543092